CLINICAL TRIAL: NCT04257383
Title: The PLAY Collaborative: Testing an Implementation Strategy for Scaling Out Evidence-Based ECD Home-Visiting in Rwanda
Brief Title: The Sugira Muryango PLAY Collaborative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: FXB (Unknown); Laterite (Unknown); LEGO (Unknown); Grand Challenges Canada (Other); Echidna Giving (Unknown); The ELMA Foundation (Other); InfaCare Pharmaceuticals Corporation, a Mallinckrodt Company (Industry)
Responsible Party: Principal Investigator, Theresa Betancourt, Salem Professor in Global Practice, Boston College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 001210997
Record Dates: First submitted 2020-01-30; First posted 2020-02-06 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Child Development; Parenting; Parent-Child Relations; Child Malnutrition
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: The proposed study design consists of a two-arm cluster randomized control trial (CRT), which will span approximately 36 cells in 3 districts of Rwanda to compare outcomes among VUP eligible households with at least one child birth-36 months old in the following study arms: treatment and waitlist control. For the embedded quasi experimental study, we aim to enroll 540 households. These households will be assessed at baseline (pre-intervention), midline (post-intervention) and endline (12-months follow-up).
Who Masked: Outcomes Assessor
Masking Description: Our study works with Laterite to oversee data collection in the field. Laterite enumerators are blind to study condition and therefore do not know which study arm participants have been clustered and randomized into.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Families in the treatment cells will receive the Sugira Muryango treatment immediately after household identification and enrollment.
  Interventions: Other: Sugira Muryango
- Waitlist Control (Experimental): Families in the control cells will receive the Sugira Muryango treatment following the completion of the 12-month follow up on the original treatment group.
  Interventions: Other: Sugira Muryango

INTERVENTIONS:
Other: Sugira Muryango — Strong Families, Thriving Children "Sugira Muryango" is a home-visiting intervention that empowers low-income families enrolled in Rwanda's social protection system to support early childhood development and healthy family functioning.

SUMMARY:
The Research Program on Children and Adversity (RPCA) has successfully grown its evidence-based home-visiting program-Sugira Muryango (SM)-in Rwanda, as policies and programs aligned with the Rwandan social protection system have evolved. The current study submission seeks to test an evidence-based implementation strategy, the PLAY Collaborative, to engage local stakeholders and frontline providers and supervisors to ensure quality improvement and sustainability of Sugira Muryango and to repeat our previous intervention to include Ubudehe 1 families with children 0-36 months in Nyanza, Ngoma, and Rubavu Districts in Rwanda.

DETAILED DESCRIPTION:
The Research Program on Children and Adversity (RPCA) has successfully grown its evidence-based home-visiting program-Sugira Muryango-in Rwanda, as early childhood development (ECD) policies and programs have evolved. The combination of ECD commitment by the government and the proven Sugira Muryango intervention creates an ideal environment for further collaboration between RPCA and families at-risk of interpersonal violence, malnutrition, and other factors crucial to successful development of children. Sugira Muryango was designed as a complement to other center and community-based ECD interventions in Rwanda that may not adequately address issues such as limited stimulation in the home, hygiene, nutrition, father engagement, and violence in the home which is more prevalent among families living in extreme poverty.

Sugira Muryango is a home-visiting model to support playful parenting, father engagement, improved nutrition, care seeking and family functioning-to promote ECD, positive parent-child relationships, and healthy child development. The intervention (a) builds playful parenting skills and improves knowledge of ECD to create a safe, stimulating and nourishing environment for the growth of young children with a focus on nutrition, health and hygiene promotion; (b) coaches parents of young children in "serve and return" interactions and playful parenting; (c) develops a "family narrative" to build hope and highlight sources of resilience for addressing challenges and reducing risk of violence; (d) strengthens problem-solving skills as well as the navigation of formal and informal community resources; and, (e) builds skills in parental emotion regulation and alternatives to harsh punishment. Sugira Muryango integrates these core components, informed by the WHO Care for Child Development package, into 12 modules and two booster/follow-up sessions. The 60-90 minute modules are delivered weekly over 3-4 months by well-trained lay interventionists embedded in the community referred to as IZUs.

The Sugira Muryango intervention has been demonstrated as clinically effective due to its theory of change, its evidence-based curriculum, and its implementation science approach. To date, RPCA's implementation science strategies have focused on: 1) determining fidelity to curriculum content and delivery and developing strategies for quality improvement; 2) evaluating how features of program delivery moderate or mediate outcomes on children and families; and 3) identifying evidence-based practices pertaining to delivery, supervision and monitoring to support a systems level scaling-up of the program. Sustainment and scaling of Sugira Muryango requires strong local buy-in and government commitment. We plan to achieve this by evaluating a new implementation science strategy-a Collaborative Team Approach (CTA), drawn from evidence-based practices in implementation science described in this project as the "PLAY Collaborative". A key feature of the PLAY Collaborative to transition the evidence-based Sugira Muryango to ownership by local stakeholders is the development of a cross-site Seed Team that will assume a leadership role in ongoing training, supervision and fidelity across a regional set of IZU interventionists. As the in-country Sugira Muryango expert, with a strong presence in our target districts, François Xavier Bagnoud (FXB)-Rwanda (hereafter FXB) will staff and lead the development and activities of the Seed Team. FXB-Rwanda has been awarded a grant from Grand Challenges Canada to start the development of the Seed Team in Nyanza district, so it will be mature and well developed to expand to all three districts under the LEGO Foundation Hybrid Type II Implementation-Effectiveness Trial. In the PLAY Collaborative strategy being evaluated therein, the Seed Team comprising Sugira Muryango experts with ECD and family violence prevention experience, will be employed by FXB and physically based near and linked to IZUs at the village level. The Seed Team will work across our three target districts to oversee Sugira Muryango delivery while establishing regional teams of IZU interventionists, Cell Coordinators and Sector Associate Trainers to embed the SM practice in the community.

By developing local expertise through regional collaborative teams, and a Seed Team that shifts ownership to local partners for training and ongoing supervision, cross-site learning, dissemination and sustainability are enhanced. The PLAY Collaborative is modeled after the Interagency Collaborative Team model utilized by Dr. Gregory Aarons in scaling up the SafeCare intervention for families involved in or at-risk for involvement in the child welfare system in the United States. Through this work, collaboration emerged as a key element for the implementation and sustainment of evidence-based practices into established service delivery systems. Within the PLAY Collaborative, collaboration primarily involves in-country Sugira Muryango experts (FXB), ECD stakeholders (NCC, NECDP, MIGEPROF), Sector Associate Trainers, Cell Mentors, and service providers (IZU interventionists). This model is uniquely aligned to sustain and scale the evidence-based SM ECD home-visiting intervention as reliance on remote expertise in low resource settings is neither feasible nor sustainable.

Two main activities will be conducted:

1. To replicate the Sugira Muryango intervention while expanding the target population and the children's age, to all Ubudehe 1 families with children between birth and 36 months in Nyanza, Ngoma, and Rubavu districts.
2. To Evaluate the implementation strategy of the PLAY collaborative and its relation to Intervention effectiveness.

Our specific hypotheses are as follows:

1. Intervention effectiveness:

   1. The updated Sugira Muryango intervention, delivered by a government-supported community volunteer workforce, will lead to improvements in responsive parent-child relationships, improved child development and reduced violence.
   2. The updated Sugira Muryango intervention will lead to improvements in caregiver behaviors that support child health including increased care seeking for illness, improved hygiene, and improved dietary diversity as well as improvements in observed child health outcomes related to child growth and illness.
2. Implementation via the Play Collaborative:

   1. Engagement and buy-in of the PLAY Collaborative will strengthen dissemination and implementation of Sugira Muryango.
   2. High fidelity to Sugira Muryango core components will enhance Sugira Muryango clinical effectiveness and improve caregiver and child outcomes.
   3. Implementation science constructs related to acceptability, feasibility, and appropriateness will be strongly and positively correlated with program satisfaction.

The effectiveness trial to evaluate the expanded Sugira Muryango program delivered within the PLAY collaborative (which targets 10,000 households across three study districts) will utilize a Hybrid Type 2 Effectiveness-Implementation study design. This design blends components of a clinical effectiveness trial with implementation science research methodology (Curran et. al, 2012). The blending of these two lines of research has several advantages over pursuing each line of research independently including more rapid translational gains, more effective implementation strategies, and more useful information for decision makers. This Hybrid Type 2 Effectiveness-Implementation Design trial will utilize the EPIS conceptual model which guides the anticipation, identification, and response to common issues when transitioning evidence-based practices to larger delivery systems such as those in the public sector where they can have the most impact.

A quasi-experitmental design with randomization at the village level will be used such that each village will either receive the treatment or care as usual, which will help in avoiding the risk of diffusion of the treatment (i.e., treatment families sharing practices learned with others who did not receive the treatment). Both quantitative and qualitative data will be collected in three timepoints (baseline, post-intervention, and 12-months follow-up) by local research assistants blind to site and family condition assignments to investigate implementation processes and impact of the Sugira Muryango intervention at multiple levels: family level, interventionist level, supervisor level, and district level.

ELIGIBILITY:
Inclusion Criteria:

Household inclusion criteria: Participants must be the primary caregiver to a child between birth and 36 months. Caregivers must live in the same household as the child and must be the child's legal guardian. Legal guardians may be parents, aunts, uncles, grandparents, or foster parents. Participants must be categorized as Ubudehe 1 under the socio-economic categorization of households from LODA.

Government Official inclusion criteria: Government officials must be located at the Village, Cell, Sector and/or District level and must participate in the 1-day ECD training. Government officials must also agree to participate in the PLAY Collaborative activities throughout the course of program delivery.

IZU interventionist inclusion criteria: IZUs must be a part of the Inshuti z'Umuryango/Friends of the Family program, must be over the age of 18, and must be literate in Kinyarwanda.

Cell Level IZU Mentor inclusion criteria: Cell Level IZU Coordinators must be situated at the Cell Level and able to supervise at least 12 IZU interventionists, they must be over 18 years of age, and must be literate in Kinyarwanda.

Exclusion Criteria:

Household exclusion criteria: Potential participants will be excluded if they do not meet the inclusion criteria above, are experiencing an active crisis (e.g., psychosis), or have severe cognitive impairments which preclude their ability to speak to the research questions/assessments under scrutiny.

Government Official exclusion criteria: Government officials will be excluded from participation in the PLAY Collaborative if they are not located at the Cell, Sector or District level and if they are unable to meet the demands of participation in the PLAY Collaborative.

IZU interventionist exclusion criteria: IZUs will be excluded from participation if they do not meet the inclusion criteria above and if they are unable to meet the demands of delivering the Sugira Muryango program.

Cell Level IZU Mentor exclusion criteria: Cell Level IZU Coordinators will be excluded if they do not meet the inclusion criteria above or are unable to meet the demands of supporting the delivery of the Sugira Muryango program.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1333 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Home Observation for Measurement of the Environment (HOME) Inventory | baseline, 4-months, 16-months
  The HOME is a 43-item survey to assess responsive caregiving. The HOME combines observation of parenting behaviors and household conditions with caregiver report. Items are summed to derive a total score with a minimum score of 0 and a maximum score of 43. Higher home scores indicate higher levels of responsive caregiving. Baseline will provide a baseline assessment of responsive caregiving while follow-up assessments will assess change over time.
Observation of Mother-Child Interaction (OMCI) | baseline, 4-months, 16-months
  The OMCI assesses responsive caregiving via a five-minute interaction that is scored according to published guidelines. The maximum OMCI score is 57 (minimum= 0) with higher scores indicating higher levels of responsive caregiving. Baseline will provide a baseline assessment of responsive caregiving while follow-up assessments will assess change over time.
UNICEF MICS Family Care Indicators (FCI) | baseline, 4-months, 16-months
  The UNICEF MICS Family Care Indicators is a cumulative score of caregivers' self-reported engagement in stimulating activities with the child during the prior three days. The maximum score is 6 (minimum score=0) with higher scores indicating higher levels of caregiver engagement in stimulating activities. Baseline will provide a baseline assessment of caregiver engagement while follow-up assessments will assess change over time.
Dissemination and Implementation Measure (D&I) | baseline and 4-months
  This measure is administered to interventionists, households, and organizations. It assess key implementation science domains related to buy-in, acceptability, feasibility, and appropriateness. Items are scored on a 4-point Likert scale (0-3) with higher scores indicating higher buy-in, acceptability, feasibility, etc. Baseline will provide a baseline assessment of these constructs while follow-up assessments will assess change over time.
Program Sustainability Assessment Tool (PSAT) | baseline and 4-months
  This assessment is administered to providers and organizations. It assesses sustainability of the Sugira Muryango intervention across 8 domains (environment, funding stability, partnerships, organizational capacity, program evaluation, program adaption, communication, strategic planning). The PSAT includes 40 items that are scored on a 7-point Likert scale (1-7) with higher scores indicating higher capacity for program sustainability. Baseline will provide a baseline assessment of program sustainability while follow-up assessments will assess change over time.
Malawi Development Assessment Tool (MDAT) | baseline, 4-months, 16-months
  The MDAT is an observational, task-based measure used to asses child development across domain of gross motor, fine motor, language and socio-emotional development. Standardization of score is done relative to data from the SHINE study from Malawi provided by the MDAT team. Baseline will provide a baseline assessment of child development while follow-up assessments will assess change over time.
Ages and Stages Questionnaire-3 (ASQ-3) | baseline, 4-months, 16-months
  The ASQ uses a series of parent-completed range age-specific questionnaires designed to screen for developmental delay of children in the areas of gross motor skills, fine motor skills, communication, and problem solving. The ASQ-3 is scored using standard guidelines for standardization resulting in binary outcome variables for each domain indicating whether or not the child showed "developmental delay" vs. "no developmental delay. Baseline will provide a baseline assessment of child development while follow-up assessments will assess change over time.
UNICEF MICS: Child Discipline Module | baseline, 4-months, 16-months
  Assesses children's exposure to violent and nonviolent discipline. Exposure to violence is assessed by summing the exposures and creating a continuous score that can range from 0 to 13. Baseline will provide a baseline assessment of child discipline while follow-up assessments will assess change over time.
Rwanda Demographic Health Survey- Intimate Partner Violence | baseline, 4-months, 16-months
  Indicators from the Rwanda DHS cover topics related to perpetration and victimization of violence between intimate partners.

SECONDARY OUTCOMES:
Rwanda Demographic and Health Survey (DHS) | baseline, 4-months, 16-months
  Indicators from the Rwanda DHS cover topics related to child health, care seeking, WASH (Water, Sanitation, Hygiene), and intimate partner violence. All responses are binary (yes/no). Baseline will provide a baseline assessment of child health while follow-up assessments will assess change over time.
WHO infant and young child feeding practices | baseline, 4-months, 16-months
  This assessment assesses children's nutritional intake was assessed by parent-reported dietary diversity reflecting the number of food groups (out of 7) the child consumed in the past 24 hours. Scores are binary (yes/no) and a sum score is created to indicate dietary diversity; minimum score is 0 and a maximum score in 14. Baseline will provide a baseline assessment of dietary diversity and nutrition while follow-up assessments will assess change over time.
Child Anthropometrics | baseline, 4-months, 16-months
  Child anthropometrics are assessed by taking child's height, weight, length and a measure of the middle-upper arm circumference. Height is measured in centimeters to the nearest 0.1 cm. Weight is measured in kilograms to the nearest 1 gram. Middle upper arm circumference is measured in centimeters to the nearest 0.1 cm. Standardization is done using software provided by the World Health Organization. Baseline will provide a baseline assessment of child height/weight/growth while follow-up assessments will assess change over time.

OTHER OUTCOMES:
Hopkin's Symptom Checklist (HSCL) | baseline, 4-months, 16-months
  Assesses caregiver mental health including two subscales related to anxiety and depression. The HSCL includes 25 items scored on a 4-point Likert scale (1-4) scores can range from 1 to 100 with higher scores indicating poorer mental health. Baseline will provide a baseline assessment of caregiver mental health while follow-up assessments will assess change over time.
Difficulties in Emotion Regulation (DERS) | baseline, 4-months, 16-months
  Assesses caregiver emotion regulation. The full DERS scale includes 36 items which are scored on a 5-point Likert scale (1-5). Higher scores indicate greater difficulties in emotion regulation with a minimum score of 36 and maximum score of 180. Baseline will provide a baseline assessment of caregiver mental health (emotion dysregulation) while follow-up assessments will assess change over time.
WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) | baseline, 4-months, 16-months
  Assesses caregiver interpersonal functioning across 6 domains (cognition, mobility, self-care, getting along, life activities, participation). The WHODAS 2.0 includes 12 items scored on a 5-point Likert scale (0-4) where scores can range from 0 to 48. Higher scores indicate worse interpersonal functioning. Baseline will provide a baseline assessment of caregiver interpersonal functioning while follow-up assessments will assess change over time.
The Implementation Leadership Scale (ILS) | baseline and 4-months
  This assessment assesses a key implementation science construct regarding leadership across 4 domains (proactive leadership, knowledgeable leadership, supportive leadership, perseverant leadership). The ILS includes 12-items scored on a 5-point Likert scale (0-4) with higher scores indicating stronger leadership. Baseline will provide a baseline assessment of leadership as it regards evidence-based practice while follow-up assessments will assess change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Betancourt, Sc.D, Principal Investigator — Boston College School of Social Work
Locations (1):
- FXB Rwanda, Kigali, Rwanda

DOCUMENTS (1):
  • Study Protocol (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT04257383/Prot_001.pdf